CLINICAL TRIAL: NCT06031363
Title: A Clinical Study on the Optimal Dose of Indomethacin Suppository for Preventing Post-ERCP Pancreatitis
Brief Title: The Optimal Dose of Indomethacin Suppository for Preventing Post-ERCP Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Rui Li, Chief of the Department of Gastroenterology, The First Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023004
Record Dates: First submitted 2023-09-02; First posted 2023-09-11 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Pancreatitis; Cholangiopancreatography, Endoscopic Retrograde; Indomethacin
Keywords: Indomethacin Suppository; Post-ERCP Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Indomethacin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Regular dosage group (Active Comparator): Give indomethacin suppository 100mg anal plug immediately after operation.
  Interventions: Drug: Indomethacin Suppository
- Low dosage group (Experimental): Give indomethacin suppository 50mg anal plug immediately after operation.
  Interventions: Drug: Indomethacin Suppository
- High dosage group (Experimental): Give indomethacin suppository 150mg anal plug immediately after operation.
  Interventions: Drug: Indomethacin Suppository

INTERVENTIONS:
Drug: Indomethacin Suppository — Patients in the regular dose group are given indomethacin suppository 100 mg anal plug immediately after operation, patients in the low dose group are given indomethacin suppository 50 mg anal plug immediately after operation, and patients in the high dose group are given indomethacin suppository 150 mg anal plug immediately after operation.
  Other Names: Indomethacin

SUMMARY:
This study is a single-center, randomized, single-blind, parallel controlled clinical study to explore the optimal dose of postoperative indomethacin suppository for the prevention of post-ERCP pancreatitis. The purpose of this study is to explore the optimal dosage of indomethacin suppository for PEP prevention, to study the control effect of indomethacin on hyperamylaseemia, and to further explore the group of patients who benefit most from this therapy.

DETAILED DESCRIPTION:
This is a single-centre, randomized, single-blind, parallel-controlled designed clinical study to explore the optimal dose of postoperative indomethacin suppository for the prevention of post-ERCP pancreatitis. The study will enroll 192 patients who undergo ERCP in the Department of Gastroenterology of the First Affiliated Hospital of Soochow University from November 2022 to October 2023, and they will be randomly assigned to 3 groups of 64 each according to the date of surgery and hospitalisation number in a random number list formed by SPSS software.

ELIGIBILITY:
Inclusion Criteria:

* According to the "Chinese ERCP Guidelines (2018 Edition)", patients with various biliary and pancreatic diseases who have indications for ERCP examination and treatment, who are at least 18 years old and have no contraindications, and who can tolerate the examination;
* Preoperative blood coagulation function, liver and kidney function indicators are in the normal range;
* The patients agreed to participate in this experiment, signed the informed consent form, and was approved by the hospital ethics committee.

Exclusion Criteria:

* Contraindications to indomethacin and other NSAIDs: such as allergy to indomethacin, severe heart failure, active peptic ulcer/bleeding, perioperative period of coronary artery bypass surgery, etc.;
* There are severe cardiovascular and cerebrovascular diseases, respiratory insufficiency and coagulation dysfunction, etc., and cannot tolerate ERCP examination;
* Those who have recently used indomethacin and other non-steroidal anti-infective drugs;
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
serum amylase concentration | before operation, 3 hours after operation, 24 hours after operation, 48 hours after operation
  blood test

SECONDARY OUTCOMES:
incidence of post-ERCP pancreatitis | 3rd day after operation
  number of people with PEP in each group / total number of people in each group
incidence of hyperamylaseemia | 3rd day after operation
  number of people with postoperative hyperamylaseemia in each group / total number of people in each group
incidence of indomethacin adverse reaction events | 3rd day after operation
  number of indomethacin-related adverse events in each group / total number of people in each group

CONTACTS AND LOCATIONS:
Overall Officials: Rui Li, Dr., Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China